CLINICAL TRIAL: NCT04507464
Title: A Physical Activity Program to Disrupt Sedentary Time in Older Latinos
Acronym: PAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ulf G. Bronas, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0739; 2P30AG022849-16 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Sedentary Behavior; Cognitive Impairment
Keywords: Sedentary Behavior; Physical Activity; Cognitive Health; Older Adults; Latinos
MeSH Terms: conditions — Sedentary Behavior; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized, controlled trial of a 6-week intervention for feasibility. Outcome measures will be obtained at baseline and at 6-weeks. Behavior choices and preference data will be continuously captured during the intervention. We will randomize 80 older Latinos from the Chicago Latino community to either an ecological momentary intervention using fitbits (n=40) or to physical activity guidelines (n=40).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ecological Momentary Intervention (Experimental): Participants will receive real time physical activity notifications via a wearable activity tracker and smartphone application.
  Interventions: Behavioral: Ecological Momentary Intervention
- Physical Activity Guidelines (No Intervention): Participants will be sent general guidelines for disruption of sedentary time.

INTERVENTIONS:
Behavioral: Ecological Momentary Intervention — Participants will wear a Fitbit that has been programmed to deliver a notification (a buzz) when activity has ceased for more than 10 minutes. They will receive suggestions on their Illumivu mEMA smartphone app on how to replace sitting time with PA such as standing up 5 times or taking 20 steps, or even performing a short (20 seconds) preferred dance routine. Fitbit data will be captured in real-time via the iCardia platform. Participants will receive reminders from their smartphones to enter real-time feedback on activity options selected and how successful they were in adopting the option. These data will allow tracking of underlying preferences for behaviors and to tailor the program accordingly.
  Other Names: Illumivu mEMA
  Arms: Ecological Momentary Intervention

SUMMARY:
To test the feasibility of an intervention designed to replace sedentary time with physical activity in older Latinos, delivered in their homes to improve cognitive function and brain connectivity.

DETAILED DESCRIPTION:
After being informed of the study and potential risks, all patients giving informed consent will undergo a focused phone interviews, followed by screening to determine eligibility. Participants that meet inclusion criteria will undergo baseline cognitive function testing via video (following NIH toolbox guidelines for remote cognitive function assessment), followed by a one week measurement of sedentary time using a physical activity monitor (actigraphy). At week 0, participants will be randomized into either a physical activity group to break up sedentary time or activity guidelines only in a 1:1 ratio. Follow up occurs at 6 weeks using the same measures as baseline.

ELIGIBILITY:
Inclusion Criteria:

* no history of major head trauma
* ownership of a smartphone
* ability to make video calls

Exclusion Criteria:

* Requires assistive ambulation;
* Unstable angina,
* Claudication
* severe arthritis,
* extreme dyspnea on exertion,
* Class III-IV heart failure;
* Current uncontrolled sustained arrhythmias,
* severe/symptomatic aortic or mitral stenosis,
* hypertrophic obstructive cardiomyopathy,
* severe pulmonary hypertension,
* active myocarditis/pericarditis,
* thrombophlebitis,
* recent systemic/pulmonary embolus (within 3 months);
* Revascularization procedures within the previous 6 months;
* Pregnancy

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf G Bronas, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Bronas UG, Marquez DX, Fritschi C, Petrarca K, Kitsiou S, Ajilore O, Tintle N. Ecological Momentary Intervention to Replace Sedentary Time With Physical Activity to Improve Executive Function in Midlife and Older Latino Adults: Pilot Randomized Controlled Trial. J Med Internet Res. 2024 Sep 5;26:e55079. doi: 10.2196/55079. PMID 39235836

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Started | 20 | 19
Completed | 19 | 19
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (4.99) | 62.16 (6.57) | 61 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 19 | 39
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Sedentary Bouts
Description: Change in number of bouts of sedentary activity at 6 weeks from baseline. One sedentary bout is defined as a 10 minute bout or longer where the activity count is less than 99 counts per minute.
  Sedentary Bout Parameters Minimum Length: 10 Minutes Minimum Count Value: 0 Counts Per Minute Maximum Count Value: 99 Counts Per Minute
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: Sedentary bouts
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
Sedentary bouts | -11.58 (22.02) | -2.47 (28.06)

2. Primary Outcome: Time in Sedentary Bouts
Description: Change from baseline to 6 weeks in minutes spent in sedentary bouts
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
Minutes | -347.7 (484.98) | -27.53 (811.07)

3. Secondary Outcome: Trail Making Test A
Description: Measure of pschycomotor speed. Subjects connect a series of encircled numbers in numerical order. The score is the time in seconds it takes the subject to complete the test. A lower score/time is better. Outcome is change in time to completion of TMT-A in seconds from baseline to 6 weeks.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
Seconds | .43 (1.27) | .31 (1.73)

4. Secondary Outcome: Trail Making Test B
Description: Measure of executive function. Subjects connect encircled numbers and letters in numerical and alphabetical order, alternating between the numbers and letters. Score is the time in seconds it takes the subject to complete the test. A lower score/time is better. Outcome is change from baseline to 6 weeks in seconds. Lower time is better.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
Seconds | -35.26 (60.35) | 7.19 (46)

5. Secondary Outcome: Picture Vocabulary Test
Description: A measure of general vocabulary knowledge and is considered to be a strong measure of crystallized abilities (those abilities that are more dependent upon past learning experiences and are relatively consistent across the adult life span). The respondent is presented with an audio recording of a word and four photographic images on the iPad screen, and is asked to select the picture that most closely matches the meaning of the word. This is repeated over 4 minutes. A theta score is very similar to a z-score, which is a statistic with a mean of zero and a standard deviation of one. A higher score is better
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
score on a scale | .20 (1.49) | .25 (1.27)

6. Secondary Outcome: List Sorting
Description: The List Sorting test requires immediate recall and sequencing of different visually and orally presented stimuli (i.e., "working memory"). Pictures of different foods and animals are displayed with accompanying audio recording and written text (e.g., "elephant"), and the participant is asked to say the items back in size order from smallest to largest, first within a single dimension (either animals or foods, called 1-List) and then on two dimensions (foods, then animals, called 2-List). List Sorting is scored by summing the total number of items correctly recalled and sequenced on 1-List and 2-List, which can range from 0-26. Higher scores indicate higher levels of working memory. Change from baseline to post-test follow-up at 6-weeks is reported.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
score on a scale | 1.26 (8.7) | 5.53 (9.64)

7. Secondary Outcome: Picture Sequence
Description: A measure developed for the assessment of episodic memory. Participants are asked to recall the sequence of pictures demonstrated over two learning trials; sequence length varies from 6-18 pictures. Participants are given credit for each adjacent pair of pictures they correctly placed. The number of adjacent pairs placed correctly for each of trials 1 and 2 is converted to a theta score and a standard score is generated. Change from baseline to 6 weeks is reported. This provides a gauge of improvement or decline from one assessment to another, irrespective of demographic factors. A change in a participant's Uncorrected Standard score (or theta score) from Time 1 to Time 2 represents an absolute change in the level of performance for that individual since the previous assessment. Higher score is better.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
score on a scale | 4.26 (13.22) | 4.32 (10.73)

8. Secondary Outcome: Oral Reading Recognition Test
Description: Participant is asked to read and pronounce letters and words as accurately as possible. Administrator scores them as right or wrong (number correct words is used). This test is a measure of reading decoding skill. The Reading Test is a measure of reading decoding skill and, like vocabulary, is considered among the crystallized abilities; those abilities are generally more dependent upon past learning experiences and consistent across the adult life span. Change in Reading Uncorrected score is reported and is useful in evaluating pure change in performance from one assessment to another. Higher change in Uncorrected score for Reading would mean that the participant is able to correctly identify more difficult words on the subsequent assessment, which may indicate developmental growth or a return to a previous higher level of functioning.Change from baseline to 6 weeks is reported. A higher score is better.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: Number of correctly pronouced words
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
Number of correctly pronouced words | 6.89 (19.14) | 1 (7.58)

9. Secondary Outcome: Crystalized Cognition
Description: This composite includes the Picture Vocabulary and Reading Tests and represent an accumulated store of verbal knowledge and skills. The composite score is derived by averaging the standard scores of each of these measures, and then deriving standard scores based on this new distribution. Uncorrected standard score is generated and reported. Crystallized Cognition Composite score is considered a global assessment of individual verbal cognition. Crystallized abilities are presumed to be more dependent on experience and less on biological influences. They represent an accumulated store of verbal knowledge and skills. Higher scores indicate higher levels of functioning. Change in uncorrected standard score from baseline to 6 weeks is reported. Higher change scores indicate improved levels of functioning
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: Uncorrected standard score
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
Uncorrected standard score | 3.95 (10.46) | .95 (5.26)

10. Secondary Outcome: Auditory Verbal Learning
Description: The Rey auditory verbal learning task is a word-list learning task in which 15 unrelated words are presented orally (via audio recording) over three consecutive learning trials1. After each presentation, the participant is asked to recall as many of the words as he/she can. The Rey is scored by taking the sum of the number of words recalled across all trials (possible range is 0-45 words). The raw score is most commonly used for interpretation of the Rey test, with higher scores representing better episodic memory. Change from baseline to post-test follow-up at 6-weeks is reported.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 19
score on a scale | .26 (4.04) | .47 (5.23)

11. Secondary Outcome: Text Message Motivation.
Description: Participant reported rating on a scale from 0-10, with 0 being no motivation and 10 being the highest motivation provided by the ecological momentary intervention text messages. Assessed at 6 weeks in the intervention group only.
Time Frame: 6 weeks.
Population: EMI ratings apply to intervention group only.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 0
units on a scale | 8.7 [3 to 10] |

12. Secondary Outcome: Enjoyment of the Text Messages.
Description: Participant reported rating on a scale from 0-10, with 0 being none and 10 being the highest, reported enjoyment of the ecological momentary intervention text messages. Assessed at 6 weeks.
Time Frame: 6 weeks.
Population: Intervention group only.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 0
units on a scale | 8.8 [0 to 10] |

13. Secondary Outcome: Text Messages Helping Exercise.
Description: Participants reported rating, on a scale from 0-10 with 0 being none and 10 being the highest, of the ecological momentary intervention text messages helping them to exercise. Assessed at 6 weeks only
Time Frame: 6 weeks.
Population: Intervention group only.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 0
units on a scale | 8.9 [0 to 10] |

14. Secondary Outcome: Difficulty Understanding Text Messages
Description: Participants reported rating, on a scale from 0-10 with 0 being none and 10 being the highest, of the ecological momentary intervention text messages being difficult to understand. Assessed at 6 weeks.
Time Frame: 6 weeks
Population: Intervention group only.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 0
units on a scale | 0.9 [0 to 10] |

15. Secondary Outcome: Enjoyment of the Program.
Description: Participants reported rating, on a scale from 0-10 with 0 being none and 10 being the highest, of the enjoyment of the ecological momentary intervention.
Time Frame: 6 weeks.
Population: Intervention group only.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 0
units on a scale | 9.4 [8 to 10] |

16. Secondary Outcome: Difficulty With the FitBit.
Description: Participants reported rating, on a scale from 0-10 with 0 being none and 10 being the highest, of difficulty using the FitBit. Assessed at 6 weeks.
Time Frame: 6 weeks.
Population: Intervention group only.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
Number analyzed (Participants) | 19 | 0
units on a scale | 1.7 [0 to 10] |

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: no difference from clinical trials definitions
Arm/Group | Ecological Momentary Intervention | Physical Activity Guidelines
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT04507464/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT04507464/ICF_001.pdf